CLINICAL TRIAL: NCT03825172
Title: Evaluation Of Caudal Epidural Anatomy By Ultrasonography İn Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Pinar Kendigelen (Unknown); Ayse Cigdem Tutuncu (Other); Kaya, Guner, M.D. (Individual)
Responsible Party: Principal Investigator, Celal Kaya, resident, Istanbul University
Other Study IDs: 72109855-604.01.01-103424
Record Dates: First submitted 2019-01-24; First posted 2019-01-31 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-04

CONDITIONS: Anesthesia, Caudal; Anatomy; Ultrasonography; Pediatrics
Keywords: Caudal block; Ultrasound; Children; Regional block anatomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: Caudal Epidural Ultrasonography will be performed in patients aged between 1-24 months
  Interventions: Diagnostic Test: Caudal Epidural Ultrasonography
- Group II: Caudal Epidural Ultrasonography will be performed in patients aged between 25-48 months
  Interventions: Diagnostic Test: Caudal Epidural Ultrasonography
- Group III: Caudal Epidural Ultrasonography will be performed in patients aged between 49-84 months
  Interventions: Diagnostic Test: Caudal Epidural Ultrasonography

INTERVENTIONS:
Diagnostic Test: Caudal Epidural Ultrasonography — Ultrasonographic Measurement

SUMMARY:
Detailed study of ultrasonographic caudal epidural anatomy

DETAILED DESCRIPTION:
Caudal epidural block is one of the most common methods to provide analgesia for an infraumbilical surgery in children. Although it can be carried out safely and easily, many complications have been described so far, because of inaccurate needle injections. To perform a successful block, a good caudal epidural anatomic assessment is essential. Ultrasonography is an important tool to perform pediatric regional blocks, including caudal blocks. We believe that caudal epidural ultrasound evaluation can be an important option to decrease complications and to achieve a successful attempt; due to that we will try to describe caudal epidural ultrasound imaging and changes from one month to 84 months.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who applied for any pediatric surgery from 20 january to 20 july

Exclusion Criteria:

* Premature patients
* Patients who have any sendromic diagnosis
* Patients who have any musculoskeletal abnormalities
* Patients who have any spinal abnormalities

Ages: 1 Month to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who are admitted to operating room for any pediatric surgery
Sampling Method: Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Definition Of Dural Sac Termination Level By Ultrasonography | 5 minutes
  After general anesthesia, patient will be placed in lateral decubitus position. First, a 12 MHz lineer ultrasound transducer will be placed transversely to obtain the transverse view of sacral hiatus; in this view we will try to show two sacral cornua, sacrococcygeal ligament, posterior sacral bone and caudal epidural depth. Secondly, transducer will be turned parallel to the midline or paravertebral to obtain longitudinal view; in longitudinal view we will try to obtain the images of sacral vertebral corpuses, caudal epidural area and dural sac. We will try to determine the level of dural sac termination according to a part of vertabral corpus or an intervertebral distance.
Distance Between Dural Sac Termination Level And Placement Of Caudal Epidural Needle | 5 minutes
  Distance Between Dural Sac Termination Level And Placement Of Caudal Epidural Needle will be measured under longitudinal ultrasound view
Definition Of Average Caudal Epidural Depth By Ultrasonography | 5 minutes
  Definition of caudal epidural depth by ultrasonography will be obtained under transverse view for every patient and average value will be defined for every age group.

SECONDARY OUTCOMES:
Determination Of Sacral Cornua As An Anatomic Landmark And Confirmation By Ultrasonography | 5 minutes
  Sacral cornua will be palpated and than will be scanned under transverse ultrasound view. Also results will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Celal Kaya, MD, Principal Investigator — Istanbul University
Locations (1):
- Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided